CLINICAL TRIAL: NCT04453891
Title: Evaluating the Feasibility of Monitoring Symptomatic COVID-19 Patients, and Predicting Disease Progression Using a Validated Digital Health Program
Brief Title: Hexoskin Feasibility Study With COVID-19 Patients
Status: Withdrawn | Type: Observational
Why Stopped: Internal timeline was delayed, logistics delays
Sponsor: Nguyen Thu Ngan Trinh (Industry)
Responsible Party: Sponsor-Investigator, Nguyen Thu Ngan Trinh, Clinical Applications Specialist, Carré Technologies Inc.
Organization: Carré Technologies Inc. (Industry)
Other Study IDs: Hexoskin COVID-19 Study
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Monitoring physiological data with the Hexoskin smart shirt — Participants will be monitored using a validated biometric garment (Hexoskin smart shirt). Cardiorespiratory and activity data will be collected over a 28-day monitoring period. Participants will be invited to wear the shirt during the day and at night.

SUMMARY:
This pilot study aims to investigate the feasibility of using Hexoskin cardiorespiratory and activity data, as well as patient symptomatology, to provide an AI model for disease progression that will be at the service of the clinical team to recommend the best customized and evolving care trajectory for each patient.

DETAILED DESCRIPTION:
The following protocol proposes a mixed methods pilot study, whereby the immediate purpose is to generate quantifiable information regarding the feasibility of a virtual trial with the Hexoskin Platform, collection of data quality in COVID-19 patients, and values for algorithm construction. In essence, sixteen participants with a confirmed COVID-19 diagnosis will be invited to wear the Hexoskin biometric garment during the course of several hours per week, over a period of 28 days. In addition to the biometric data collection, participants will be invited to complete four questionnaires. The biometric data will be combined to the sociodemographic information and patient symptomatology to construct an algorithm which can accurately predict patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Minimum waist size of 24 inches, and maximum waist size of 45 inches
* Confirmed COVID-19 diagnosis from a licensed healthcare practitioner
* Permanent resident or citizen of the United States
* Access to a smartphone
* Access to a functional email
* Access to a thermometer
* Access to a measuring tape
* Experiencing at least three of the following COVID-19 symptoms (fever, cough, difficulty breathing, intense fatigue, sudden loss of smell and/or taste without nasal congestion, sore throat, headache, aching muscles, loss of appetite, diarrhea).

Exclusion Criteria:

* Hexoskin should not be used by people with allergies to the following materials: polyester, synthetic fibers. Usage must be stopped if the product causes skin irritation or rashes.
* Hexoskin should not be used by people with Pacemakers or Implantable Cardioverter-Defibrillator (ICD) devices.
* Hexoskin must not be used simultaneously with a Holter Monitor, as the equipment would interfere with the placement of the Hexoskin sensors.
* Hexoskin must not be used in an MRI machine as it contains metallic parts.
* Individuals who do not fit any of the Hexoskin Shirts sizes (Men: between 2XS - 6XL, Women: between 2XS - 4XL).
* Individuals who have a documented medical condition or illness requiring intensive medical treatment.
* Women of Childbearing Potential whom are not using effective contraceptive measures

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients aged 55 and above, and resident of any state in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of the feasibility of the Hexoskin Platform and Virtual Recruitment Process via three subjective feedback questionnaires provided to all patients enrolled in the study. | Up to six months
  Evaluating the feasibility of a virtual trial to collect physiological data with the Hexoskin Platform.
Ensure the collection of high-quality data during wake and sleep activities, registered as overall > 90% good quality cardiac data and overall > 90% good quality respiratory data per recording. | Up to six months
  Assessing the quality of the data collected with Hexoskin with the Hexoskin quality assessment channels from patients recruited during a virtual trial.
Ensure adequate patient compliance, qualified as > 75% of total recording hours completed, and > 75% of daily questionnaires completed. | Up to six months
  Determine the participant's level of compliance with study procedures of the research protocol.
Investigate the predictive power of Hexoskin physiological data, patient information and symptoms information to correctly classify patient disease progression quantified as the area under the receiver operator characteristics curve (AUC ROC > 0.70). | Up to six months
  Assessing the feasibility to use the data collected to build a predictive algorithm for the Hexoskin Remote Monitoring Platform.

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Thu Ngan Trinh, Principal Investigator — 1-888-887-2044

IPD SHARING:
Plan to Share IPD: No